CLINICAL TRIAL: NCT00344838
Title: Customized Laser Ablation: Comparing Results of LADAR Vision and VISX Platforms
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James McCulley, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: 0903-556
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Customized Laser Ablation
Keywords: LADARWave™; WaveScan Wavefront™ Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Comparison of LADAR CustomLasik and VISX Wavefront System custom laser ablation devices

SUMMARY:
To compare the results of two commercially available customized laser ablation devices.

DETAILED DESCRIPTION:
In the past few years, several custom laser ablation platforms have emerged in the marketplace but only two are currently approved by the FDA. They are the LADAR CustomLasik (Alcon: Ft. Worth, TX) and the VISX Wavefront System (VISX: Santa Clara, CA). Although both use the Hartmann-Shack wave sensing principle, there are some basic distinctions in wave capture and processing technology. Moreover, there are fundamental differences in as far as centration, registration, and ablation technology is concerned. Evaluating and comparing the results of these two systems in assorted categories of patients would help us select the appropriate laser platform for the patient.

Once a patient has been scheduled to undergo customized laser ablation, they will have a routine preoperative examination. The following tests will be gathered and evaluated by the doctor in order to determine eligibility for the treatment. If the patient qualifies for custom laser ablation, this information will also be used for the study as long as they give written consent.

Pre-operative Visit (Screening visit): Date of Visit, Patient Initials, Date of Birth, Sex, Race, Assessment of visual needs, Ocular history, History of contact lens wear, Medical history, Allergies to food and drugs, Medication, family history, Distance and Near Vision (with and without correction), Auto-refraction, Refraction, eye dominance, Keratometry, Visual Acuity, Pupil size (bright and dim lighting), Afferent Pupillary Defect (ADP), Ocular motility, Ophthalmoscopy, Cycloplegic refraction, Pachymetry, Intaocular Pressure test, Custom Vue (VISX), LADARWave (LADAR), and Schirmers testing with anesthetic. Typically, these procedures are employed as part of "standard of care" for patients who are seeking custom LASIK treatment. Furthermore, there will be two additional procedures that will be performed as "reseach" measures . These are visual acuity with an Early Treatment Diabetic Retinopathy Study (ETDRS) vision chart and contrast sensitivity.

Post-Operative visits (Day 1, Week 1, Month 1, Month 3, Month 6, and Month 12): ETDRS Visual Acuity, contrast sensitivity along with a questionnaire pertaining to the study patients visual problems and experience will be completed by the patient at week 1 and after each visit thereafter. These procedures are intended as part of research.

Additional data gathered as part of "standard of care" will include: date of visit, patient initials, visual acuity, refraction, Intraocular Pressure (discretion of physician), Custom Vue (VISX) and LADARWave. Both Custom Vue and LADAR measurements are taken at 3-month visit only!

The research project proposes to compare the results of two FDA approved laser ablation treatment methods. While both treatment modalities are considered standard of care for those who decide to perform customized laser treatment, the "comparison" is intended as part of this research project.

ELIGIBILITY:
Inclusion Criteria: Individuals of both genders, aged 18 and older, who have been scheduled to undergo customized laser ablation will be considered for this prospective study.

Exclusion Criteria: There are no exclusion criteria available for this study.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Refractive Surgery Eligible Candidates
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2003-09; Primary Completion 2015-12 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Aberration Assessment | 12 Months
  Visual Acuity aberration pre-and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: James P. McCulley, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States